CLINICAL TRIAL: NCT00400322
Title: A Randomized Double Blind Controlled Proof of Concept Study of the Efficacy and Safety of Valcyte® as an add-on Therapy in Patients With Malignant Glioblastoma With Successful Surgical Resection of at Least 90 % of the Initial Tumor and CMV Infection Demonstrated Histologically and Immunohistochemically.
Brief Title: Efficacy and Safety of Valcyte® as an add-on Therapy in Patients With Malignant Glioblastoma and Cytomegalovirus (CMV) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Cecilia Soderberg-Naucler, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MV20145; 2006-002022-29 (EudraCT Number)
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Glioblastoma Multiforme; Cytomegalovirus Infection
Keywords: glioblastoma multiforme; cytomegalovirus infection; antiviral treatment; valganciclovir
MeSH Terms: conditions — Glioblastoma; Cytomegalovirus Infections | interventions — Valganciclovir

ARMS (2):
- Valganciclovir (Active Comparator)
  Interventions: Drug: Valganciclovir (Valcyte)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Valganciclovir (Valcyte)
  Arms: Valganciclovir
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate if treatment of CMV infection by antiviral drug Valcyte (R) affects the clinical outcome of glioblastoma multiforme in patients with local CMV infection in tumor tissue. The investigators' hypothesis states that CMV infection promotes tumor development and disease progression and inhibits immune responses against the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Glioblastoma grade IV
* Cytomegalovirus detected in tumor
* At least 90% resection of tumor

Exclusion Criteria:

* Decreased kidney function
* Pregnancy
* Neutropenia
* Thrombocytopenia
* Patient not tolerating the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Tumor size | Week twelve
Tumor size | Week twenty four

SECONDARY OUTCOMES:
Disease status | 24 months
Patient survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Inti Peredo, MD, Principal Investigator — Karolinska University Hospital; Cecilia Soderberg-Naucler, MD, PhD, Study Chair — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Department of neurosurgery, Karolinska University Hospital, Solna, Stockholm County
  - Department of Oncology, Norrland University Hospital, Umeå
  - Department of Oncology, Akademiska Hospital, Uppsala